CLINICAL TRIAL: NCT02693431
Title: Impact of Art Therapy on Anxiety Identified During the Quarterly Update of Hospitalizations Among Children With Cystic Fibrosis Aged 8 to 13 - Pilot Study
Brief Title: Impact of Art Therapy on Anxiety Identified During Hospitalizations Among Children With Cystic Fibrosis Aged 8 to 13
Acronym: MUCO-ART
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0459
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional Study — Parents and children will be informed at the inclusion visit (V0) that is a normal consultation under the care of the child.
  The children included will be followed for 18 months with a maximum of 6 months without meeting art therapy sessions and 12 months with art therapy. The art therapy sessions will be scheduled during the usual consultations conducted as part of the care of children.
  At each visit, clinical, paraclinical and external factors of anxiety will be collected and anxiety of parents and children will be measured using specific questionnaires.

SUMMARY:
Currently the management of cystic fibrosis (CF) patients is mainly based on symptomatic treatments. The arrival of children in day hospital, every 2 to 3 months, is for many of them and those around them, stressful, rarely expressed, but noticeable by the care team. In line with the recommendations of the High Authority of Health, the multidisciplinary team of Resources and Skills Centre for Cystic Fibrosis (CRCM) Pediatric of Nantes University Hospital offers a therapeutic education program tailored to the needs of children with cystic fibrosis and their families . The aim is to support children and parents in the acquisition of self-care skills (knowledge and skills) and coping skills, such as managing stress and emotions . Our goal is to demonstrate that art therapy, mobilizing coping skills of the child, facilitates its expressive capabilities and reduces anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Children with CF aged 8 to 13 years as part of their monitoring at CRCM children of Nantes University Hospital
* Parents and children willing to participate in research

Non inclusion Criteria:

* Emergency consultation
* Planned move

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 27 children (and their parents) aged 8 to 13 years in 2016 with cystic fibrosis followed at CRCM children Nantes.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Changes in the overall score of children's anxiety after 4 visits including art therapy sessions compared to basal mean level of the first two visits without art therapy. | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie DAVID, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No